CLINICAL TRIAL: NCT00837330
Title: Treatment of Polypoidal Choroidal Vasculopathy With Ranibizumab(Lucentis): A Phase I/II Safety Study.
Brief Title: Ranibizumab (Lucentis) for Polypoidal Choroidal Vasculopathy
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Southeast Retina Center, Georgia (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Principal Investigator, Dennis M. Marcus, M.D., Dr. Dennis M. Marcus Principal Investigator, Southeast Retina Center, Georgia
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FVF3761s
Record Dates: First submitted 2009-02-04; First posted 2009-02-05 (Estimated); Results first posted 2014-06-23 (Estimated); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Polypoidal Choroidal Vasculopathy
Keywords: polypoidal choroidal vasculopathy; choroidal neovascularization; ranibizumab; Lucentis
MeSH Terms: conditions — Polypoidal Choroidal Vasculopathy; Choroidal Neovascularization | interventions — Ranibizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ranibizumab 0.5 mg/ 0.05 cc (Experimental): Intraocular injection of 0.5 mg/ 0.05 cc ranibizumab
  Interventions: Drug: ranibizumab 0.5 or 0.3 mg/0.05 cc
- Ranibizumab 0.3 mg/ 0.05 cc (Experimental): Intraocular injection of 0.3 mg/ 0.05 cc ranibizumab
  Interventions: Drug: ranibizumab 0.5 or 0.3 mg/0.05 cc

INTERVENTIONS:
Drug: ranibizumab 0.5 or 0.3 mg/0.05 cc — ranibizumab 0.5 or 0.3 mg/0.05 cc administered intraocularly on a monthly basis for 3 months, followed by monthly examination with the option of further ranibizumab treatment or other therapies at the discretion of the treating physician
  Other Names: Lucentis

SUMMARY:
This Phase I/II safety study is designed to investigate the safety and efficacy of ranibizumab (Lucentis) in the treatment of polypoidal choroidal vasculopathy (PCV), a potentially blinding eye disease that involves the growth of tiny, abnormal blood vessels under the retina. These abnormal blood vessels can bleed or leak fluid, causing disruption of normal retinal function and vision loss. Ranibizumab is a drug that is FDA-approved for the treatment of wet age-related macular degeneration (AMD) and is injected directly into the eye. Given the efficacy of ranibizumab in the treatment of wet AMD, and the postulated similarity between the disease mechanisms involved in both wet AMD and PCV, we believe ranibizumab will have a beneficial effect on visual function in patients with PCV.

DETAILED DESCRIPTION:
Please see above description. Phase I/II safety study; prospective, open-label, single-center, non-randomized, uncontrolled, consecutive interventional case series. Enrolled patients are >35 years old and display exudative, active polypoidal choroidal vasculopathy (PCV) in 1 eye. PCV is defined as choroidal neovascularization that displays occult characteristics on fluorescein angiography and polypoidal interconnecting vascular channels with saccular dilatations on indocyanine green angiography and/or fluorescein angiography. Eyes receive 3 consecutive, monthly intravitreal ranibizumab injections (0.5 mg or 0.3 mg/0.05 cc) followed by monthly evaluations with the option of additional intravitreal ranibizumab or alternative treatments at the discretion of the investigator. Baseline and follow-up evaluations include medical history, blood pressure, physical examination, early treatment diabetic rentinopathy study (ETDRS) best-corrected visual acuity (BCVA), intraocular pressure measurement, complete ophthalmologic examination, fundus photography, fluorescein/ indocyanine green (ICG) angiography, and optical coherence tomography (OCT).

ELIGIBILITY:
Inclusion Criteria:

* Age >35 years
* Exudative, active PCV in 1 eye.
* PCV is defined as choroidal neovascularization that displays occult characteristics on fluorescein angiography and polypoidal interconnecting vascular channels with saccular dilatations on indocyanine green angiography and/or fluorescein angiography.

Exclusion Criteria:

* Age <35 years
* Prior treatment with non-ranibizumab therapies (e.g., laser, surgery, or bevacizumab)

Min Age: 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2006-05; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dennis M. Marcus, M.D., Principal Investigator — Southeast Retina Center
Locations (1):
- Southeast Retina Center, Augusta, Georgia, United States

REFERENCES:
- [Derived] Marcus DM, Singh H, Lott MN, Singh J, Marcus MD. Intravitreal ranibizumab for polypoidal choroidal vasculopathy in non-Asian patients. Retina. 2013 Jan;33(1):35-47. doi: 10.1097/IAE.0b013e3182618be0. PMID 22990319

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Twenty subjects from one site in the United States will be enrolled. Subjects with active, exudative-PCV who have provided informed consent will be eligible. Date of first subject enrolled: May 19, 2006. Date of last subject enrolled: October 8, 2008.
Groups:
- Intraocular Injection 0.5 mg Ranibizumab: 10 patients will receive intraocular injection 0.5 mg ranibizumab
- Intraocular Injection 0.3 mg Ranibizumab: 10 patients will receive intraocular injection 0.3 mg ranibizumab
Period: Overall Study
Arm/Group | Intraocular Injection 0.5 mg Ranibizumab | Intraocular Injection 0.3 mg Ranibizumab
Started | 10 | 10
Completed | 9 | 7
Not Completed | 1 | 3
Not completed — Lost to Follow-up | 1 | 3

BASELINE CHARACTERISTICS:
Population: 10 subjects were enrolled into each of the two ranibizumab groups (0.3 mg/ 0.5 mg)
Groups:
- Ranibizumab 0.5 mg/ 0.05 cc: Intraocular injection of 0.5 mg /0.05 cc ranibizumab
- Ranibizumab 0.3 mg/ 0.05 cc: Intraocular injection of 0.3 mg /0.05 cc ranibizumab
- Total: Total of all reporting groups
Arm/Group | Ranibizumab 0.5 mg/ 0.05 cc | Ranibizumab 0.3 mg/ 0.05 cc | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 7 | 11
  >=65 years | 6 | 3 | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 64 (14) | 65 (8) | 64 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 7 | 12
  Male | 5 | 3 | 8
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: Commonly Reported and Notable Adverse Events
Description: Incidence and severity of ocular adverse events, as identified by indirect and direct examination. Examples include 30 letter loss, major subretinal hemorrhage, involving 75% or more of clinical macula (arcade to arcade), disease-related vitreous hemorrhage, injection-related endopthalmitis, retinal detachment, vitreous hemorrhage, study drug/procedure related uveitis, incidence and severity of other adverse events, as identified by physical examination, subject reporting, and changes in vital signs.
Time Frame: 2 years
Measure: Number; unit: participants
Groups:
- Ranibizumab 0.5 mg: Intraocular injection of 0.5 mg ranibizumab
- Ranibizumab 0.3 mg: Intraocular injection 0.3 mg ranibizumab
Arm/Group | Ranibizumab 0.5 mg | Ranibizumab 0.3 mg
Number analyzed (Participants) | 10 | 10
participants
  Spider webs | 1 | 2
  Eye pain, burning | 2 | 3
  Wavy Lines | 1 | 2
  Seeing Dark spots | 2 | 2
  Flashes of Light | 1 | 1
  Floaters | 4 | 1
  Worsening visual acuity | 2 | 1
  Eye irritation | 1 | 2
  Mild Vitreous Hemorrhage | 1 | 2
  Blurry vision | 2 | 3
  Eyelid swelling | 2 | 1
  Transient increased blood pressure | 0 | 2
  Injection-related pain | 2 | 3
  Injection-related eyelid swelling | 2 | 1
  Macular hole | 0 | 1
  Transient increased intraocular pressure | 0 | 1
  Chalazion | 1 | 0
  Stye | 2 | 0
  Decreased color vision | 0 | 1
  Foreign Body Sensation | 1 | 0
  Posterior Vitreous detachment | 0 | 1
  Retinal Pigment epithelial changes | 0 | 1
  Worsened Night Vision | 1 | 0
  Worsened polypoidal choroidal vasculopathy | 1 | 0
  Worsening of Cataracts | 1 | 2
  Itchy, watery eyes | 1 | 2

ADVERSE EVENTS:
Time Frame: 2 years
Groups:
- Ranibizumab 0.5 mg; Ranibizumab 0.3 mg: Intravitreal Injection of Ranibizumab 0.5 mg
Arm/Group | Ranibizumab 0.5 mg | Ranibizumab 0.3 mg
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 9/10 | 8/10
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ranibizumab 0.5 mg (N=10) | Ranibizumab 0.3 mg (N=10)
Flashes of Light (Eye disorders) | 1 (1) | 1 (1) — Subject sees flashes of light
Worsening of Cataract (Eye disorders) | 1 (1) | 2 (3)
Injection Site Pain (Eye disorders) | 2 (4) | 3 (3) — Self-reported ocular pain at injection site immediately following injection
Itchy, Watery Eyes (Eye disorders) | 1 (1) | 2 (4) — Self-reported itchy, watery eyes caused by seasonal allergies
Vitreous Hemorrhage (Eye disorders) | 1 (1) | 2 (2) — Vitreous hemorrhage identified on clinical exam
Ocular Blurriness (Eye disorders) | 2 (6) | 3 (4) — Self-reported ocular blurriness
Macular Hole (Eye disorders) | 0 (0) | 1 (2) — Macular Hole identified on clinical exam
Increased Intraocular Pressure (Eye disorders) | 0 (0) | 1 (2) — Increased Intraocular Pressure identified on exam
Retinal Pigment Epithelial Changes (Eye disorders) | 0 (0) | 1 (1) — Retinal Pigment Epithelial Changes identified on clinical exam
Chalazion (Eye disorders) | 1 (1) | 0 (0) — Chalazion identified on clinical exam
Seeing Dark Spots (Eye disorders) | 2 (3) | 2 (2) — Dark spots in vision after injection reported by subject
Floaters (Eye disorders) | 4 (4) | 1 (2) — Self-reported floaters seen in vision after injection
Worsened Visual Acuity (Eye disorders) | 2 (3) | 1 (2) — Worsened Visual Acuity identified on exam
Eyelid Swelling (Eye disorders) | 2 (2) | 1 (1) — Eyelid swelling identified on exam after injection
Foreign Body Sensation (Eye disorders) | 1 (1) | 0 (0) — Foreign Body Sensation reported in eye by patient
Stye (Eye disorders) | 2 (2) | 0 (0) — Stye identified on clinical exam
Posterior Vitreous Detachment (Eye disorders) | 0 (0) | 1 (1) — Posterior Vitreous Detachment identified on clinical exam
Spider Webs in Vision (Eye disorders) | 1 (1) | 2 (3) — Spider webs in vision reported by subject after injection
Wavy Lines (Eye disorders) | 1 (1) | 2 (2) — Self reported wavy lines in vision
Worsened PCV (Eye disorders) | 1 (1) | 0 (0) — Active PCV identified on clinical exam
Worsened Night Vision (Eye disorders) | 1 (1) | 0 (0) — Worsened vision at night time reported by subject
Decreased color vision (Eye disorders) | 0 (0) | 1 (1) — Subject reported decreased ability to see colors

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes